CLINICAL TRIAL: NCT04120701
Title: CIRCULATING TUMOR DNA BASED DECISION FOR ADJUVANT TREATMENT IN COLON CANCER STAGE II
Acronym: CIRCULATE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 70 - CIRCULATE
Record Dates: First submitted 2019-10-08; First posted 2019-10-09 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Patients With Resected Stage II Colon Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Chemotherapy (Experimental)
  Interventions: Drug: mFOLFOX6
- Follow-up within the study (No Intervention)
- Follow-up outside the study (No Intervention)

INTERVENTIONS:
Drug: mFOLFOX6 — Patients receive adjuvant chemotherapy every 2 weeks during 6 months: FOLFOX6m (5-FU, leucovorin and oxaliplatin).
  Arms: Chemotherapy

SUMMARY:
The objective of CIRCULATE trial is to improve care of patients after colon tumor surgery, based on an innovative marker: circulating tumor DNA.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent obtained prior to any study specific procedures
* Age ≥ 18 years and ≤ 75 years
* Histologically confirmed stage II colon and high rectum adenocarcinoma excluding low and medium rectal cancers (tumor location ≥ 12 cm from the anal verge by endoscopy and/or above the peritoneal reflection at surgery are still eligible), without gross or microscopic evidence of residual disease after surgery with curative intent. Pathology report must be faxed to CRGA just after patient's randomization.
* At least 12 lymph nodes analyzed
* Patient with MSI + tumors can be included
* All patients must have been discussed in multidisciplinary meetings with a decision of not performing adjuvant chemotherapy
* No metastatic disease on CT-Scan and/or liver MRI done within 3 months before randomization.
* Randomization planned up to 7 weeks after curative R0 resection
* WHO performance Status < 2
* No prior chemotherapy for colo-rectal cancer
* No prior abdominal or pelvic irradiation for colo-rectal cancer
* Life expectancy of ≥ 5 years
* Adequate haematological function: with neutrophils ≥ 1,500 /mm3, platelet count ≥ 100,000/mm3, hemoglobin ≥ 9 g/dL (5,6 mmol/l)
* Total bilirubin ≤ 1.5 x ULN (upper limit of normal)
* ASAT and ALAT ≤ 2.5 x ULN
* Alkaline phosphatase ≤ 2.5 x ULN
* Serum creatinine ≤ 120 µmol/L or creatinine clearance ≥50 ml/min according MDRD (Modification of Diet in Renal Disease)
* Carcinoembryogenic antigen (CEA) ≤ 1.5 x ULN after surgery (during screening period)
* Negative pregnancy test for registration(for women of childbearing age)
* Patient affiliated to a social security system

Exclusion Criteria:

* T4b tumors
* Peripheral neuropathy > grade 1
* Comorbidity influencing the 5 year patients' survival including clinically relevant cardiovascular disease,
* Ischemic myocardial infarction in the last year and/or unstable ischemic cardiopathy,
* Participation to another interventional study for postoperative therapy
* Partial or complete DPD deficiency
* Legal incapacity or physical, psychological social or geographical status interfering with the patient's ability to sign the informed consent or to finish the study
* Medical history of other concomitant or previous malignant disease, except adequately treated in situ carcinoma of the uterine cervix, basal or squamous cell carcinoma of the skin, or cancer in complete remission for ≥ 5 years,
* Lack of effective contraception in patients (men and/or women) of childbearing age, pregnant or breastfeeding women. Women of childbearing potential should agree to use a method of contraception during treatment of the trial and at least 4 months after discontinuation of oxaliplatin therapy and at least 30 days after discontinuation of 5-fluorouracil. Men must agree to use a method of contraception during treatment and at least 6 months after stopping oxaliplatin therapy and at least 3 months after stopping 5-fluorouracil.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1980 (Estimated)
Dates: Start 2020-01-17 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
3-year Disease-Free Survival in ctDNA positive patients | 3-years

CONTACTS AND LOCATIONS:
Locations (1):
- Fédération Francophone de Cancérologie Digestive, Dijon, France